CLINICAL TRIAL: NCT02185989
Title: Early Rehabilitation Combining Daily Electrical Muscle Stimulation and Early Bedside Cycling Exercise, Compared to Early Standard Rehabilitation. A Randomized, Assessor-blinded, Single-center Study in Intensive Care Patients.
Brief Title: Electrical Muscle Stimulation and Bicycling Combined to Early Standard Rehabilitation in the ICU
Acronym: PROMOREA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHRO 2014-001; ID RCB : 2014-A00566-41 (Other: ANSM; Ministry of Health ; French government)
Record Dates: First submitted 2014-07-04; First posted 2014-07-10 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: ICU-acquired Muscle Weakness
Keywords: Critical Illness/*rehabilitation; Humans; *Intensive Care Units; Muscle Weakness/diagnosis/*etiology/physiopathology/prevention & control; Polyneuropathies/diagnosis/*etiology/physiopathology
MeSH Terms: conditions — Muscle Weakness; Polyneuropathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrical muscle stimulation and bicycling (Active Comparator): Patients will undergo early electrical stimulation of the quadriceps and early leg bicycling in addition to routine care (which comprises early standard mobilization)
  Interventions: Other: Early electrical stimulation and early leg bicycling added to early standard rehabilitation
- Standard early passive/active rehabilitation (No Intervention): In this control group, patients will undergo routine care that comprises standard early passive/active rehabilitation delivered by physiotherapist with the assistance of ICU nurses

INTERVENTIONS:
Other: Early electrical stimulation and early leg bicycling added to early standard rehabilitation
  Arms: Electrical muscle stimulation and bicycling

SUMMARY:
Early mobilization (from the first day if possible), first passive and then passive and active, is recommended for critically ill patients in whom it reduces the duration of mechanical ventilation, the length of hospital stay, improves functional status, muscle strength and quality of life after hospital discharge. The early addition of leg bicycling on a cyclo-ergometer is now part of common practice in the ICU. It can preserve or improve muscle strength and further increase the beneficial effects of early mobilization. Electrical muscle stimulation of the quadriceps, is practiced in some intensive care units, and it should, in theory, also through an improvement of muscle strength, increase the beneficial effects of early mobilization.

We hypothesized that early quadriceps electrical stimulation and early work on a cyclo-ergometer associated with a standard protocol of early passive/active mobilization in the ICU may improve muscle function and reduce the duration of mechanical ventilation, length of stay, the number of readmissions and improve the quality of life in the mid term in critically ill patients, as compared to a conventional protocol of early passive/active mobilization.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 yrs
* expected length of stay in the ICU higher than 72 hours
* motor autonomy sufficient for independent ambulation (ass assessed by patient/family/familial practitioner interview

Exclusion Criteria:

* Opposition expressed by the patient, his/her legal representative or a member of his/her family
* Pregnant woman
* Resuscitated cardiac arrest before inclusion
* Patient carrying a pacemaker or an implantable defibrillator
* Patient under extracorporeal membrane oxygenation
* Severe acute cerebral disease requiring deep sedation
* Brain death
* Guillain-Barré syndrome
* Myasthenia gravis
* Known Dementia than can affect the main endpoint assessment
* Deep venous thrombosis or pulmonary embolism treated for less than 48 hours, or floating clot in femoral, iliac of inferior vena cava veins
* Unstable traumatic injuries of the spine
* Severe skin disease or surgical reasons that either prevent performing electrostimulation or bicycling in the next 2 days, or prevent patient's verticalization or transfer to chair in the next 5 days
* Amputation of a lower limb at the trans-metatarsal level or higher
* Inclusion in another interventional study with muscle strength assessment as the primary endpoint
* Moribund patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2016-11-24 (Actual)

PRIMARY OUTCOMES:
Global muscle strength assessed by the MRC (Medical research Council, 1978) score | on the day of ICU discharge (+/- 1 day)
  Global muscle strength assessed by the MRC (Medical research Council, 1978) score on the day of ICU discharge (+/- 1 day) in all enrolled patients discharged alive from the ICU. This evaluation will be conducted by a physiotherapist blinded to the randomization group

SECONDARY OUTCOMES:
Changes in thickness of the rectus femoris muscle of each thigh | from inclusion to ICU discharge (+ / - 1 day)
  Changes in thickness of the rectus femoris muscle of each thigh, as measured by ultrasound imaging, between inclusion and ICU discharge (+ / - 1 day).
Frequency of delirium in the ICU. | During ICU stay
  Delirium is defined by the CAM-ICU scale (Ely CCM 2001 Ely JAMA 2001).
Quality of life | 6 months after ICU discharge
  Quality of life 6 months after ICU discharge assessed by the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Boulain, MD, Principal Investigator — Centre Hospitalier Régional d'Orléans, France
Locations (1):
- Centre Hospitalier Régional d'Orléans, Orléans, France

REFERENCES:
- [Derived] Fossat G, Baudin F, Courtes L, Bobet S, Dupont A, Bretagnol A, Benzekri-Lefevre D, Kamel T, Muller G, Bercault N, Barbier F, Runge I, Nay MA, Skarzynski M, Mathonnet A, Boulain T. Effect of In-Bed Leg Cycling and Electrical Stimulation of the Quadriceps on Global Muscle Strength in Critically Ill Adults: A Randomized Clinical Trial. JAMA. 2018 Jul 24;320(4):368-378. doi: 10.1001/jama.2018.9592. PMID 30043066